CLINICAL TRIAL: NCT06687707
Title: EVALUATION OF PROFESSIONAL ATTITUDE, JOB SATISFACTION AND BURNOUT LEVELS OF PHYSIOTHERAPISTS
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Alper Kemal Gürbüz, Research Asistant, Kırıkkale University
Other Study IDs: Gurbuz06
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Health Personnel Attitude; Job Satisfaction; Professional Burnout
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiotherapist
  Interventions: Other: Attitude Scale towards Physiotherapy Profession; Other: Minnesota Job Satisfaction Scale; Other: Maslach Burnout Scale

INTERVENTIONS:
Other: Attitude Scale towards Physiotherapy Profession — It is a questionnaire that evaluates the attitudes of physiotherapists with 35 questions under 3 headings: professional satisfaction, qualifications required by the profession, and concerns about the profession. It was developed in 2018 by Begümhan Turhan. In this scale, which is a Likert-type questionnaire, each question is scored between 0 and 5 points. The minimum score that can be obtained from the scale is 35 and the maximum score is 175. A high score indicates that physiotherapists have a positive attitude towards their profession
Other: Minnesota Job Satisfaction Scale — It is a 20-item Likert-type questionnaire. Scores less than 3 points indicate low job satisfaction. Turkish validity and reliability studies were conducted. The validity and reliability study in Turkey was conducted by Baycan and the Cronbach's alpha value of the scale was found to be 0.77. It is a tool consisting of 20 items with features that reveal internal and external job satisfaction factors. The neutral satisfaction score of the scale is 3. If the score obtained from the scale is less than 3, job satisfaction is considered low, and if it is greater than 3, job satisfaction is considered high.
Other: Maslach Burnout Scale — The Burnout Inventory, which was developed by Maslach and Jackson (1981) and introduced to the literature under Maslach's name, is a seven-point Likert-type scale and consists of a total of 22 items and three subscales. Among these subscales, emotional exhaustion subscale consists of 9 items, depersonalisation subscale consists of 5 items and personal accomplishment subscale consists of 8 items. Scale items are scored as '1 never' and '7 always'. The Turkish validity and reliability of the questionnaire was conducted by Burhan Çapri. It is a 5-point Likert-type scale measured with 0: never 4: always options. High scores are expected

SUMMARY:
Our study was planned to investigate the professional attitudes and satisfaction levels of physiotherapists.

It has affected each professional group in different ways. The effects on health workers such as doctors and nurses have been studied in various studies.

However, there are no studies on the effects on physiotherapists. After individuals start their profession In time, they develop an attitude towards their profession through cognitive and emotional orientations. Level of interest in the profession, academic education activities related to the profession, working places, the institution where they work, the level of professional satisfaction of physiotherapists determinant factors of the disease. This study is a prospective questionnaire study. A questionnaire created through Google forms The survey will be conducted by reaching physiotherapists. The survey will start after ethics commission permission is obtained. Age, gender of individuals, year of graduation, level of education, marital status, institution, position/task, occupation of the manager of the organisation, most difficult patient group, the professional field he/she feels most deficient in, the number of training-courses he/she has taken related to the profession after graduation, after graduation The number of congresses-seminars-symposiums related to the profession, the status of following current developments will be questioned; attitude towards physiotherapy profession scale, Minnesota job satisfaction scale, motivation feedback questionnaire, Maslach burnout scale will be applied 1 time. The data will be analysed with SPSS 21.0 (SPSS Inc., Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

To have a bachelor's degree in Physiotherapy and Rehabilitation To be actively practicing the profession of physiotherapist in any institution

Exclusion Criteria:

Graduated but not working as a physiotherapist.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include individuals who graduated from the department of physiotherapy and rehabilitation and are actively working as physiotherapists. Individuals will be informed about the study and will be asked to answer the questionnaires via Google forms. Individuals will be asked to approve the consent form.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Scale | 5 minute
  Total score is calculated and used in the analysis

SECONDARY OUTCOMES:
Minnesota Job Satisfaction Scale | 5 minute
  Total score is calculated and used in the analysis
Attitude Scale Towards Physiotherapy Profession | 5 minute
  Total score is calculated and used in the analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes